CLINICAL TRIAL: NCT01439425
Title: Weight Reduction Alone May Not be Sufficient to Maintain Disease Remission in Obese Patients With Psoriasis: a Randomized, Investigator-blinded Study
Brief Title: Weight Reduction Alone May Not be Sufficient to Maintain Disease Remission in Obese Patients With Psoriasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Micol Del Giglio, Resercher, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WRP
Record Dates: First submitted 2011-08-31; First posted 2011-09-23 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Psoriasis
Keywords: psoriasis; obesity; body mass index; disease remission; diet
MeSH Terms: conditions — Psoriasis; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- weight loss (Experimental): balanced diet scheme, based on a caloric intake reduction related to BMI and sex (range: 1200-1500 kcal/d for women, 1300-1600 kcal/d for men).
  Interventions: Behavioral: Weight Loss

INTERVENTIONS:
Behavioral: Weight Loss — The low-calorie diet was designed to achieve a loss of 5-10% of initial body weight. The caloric restriction was 500 kcal below the resting energy expenditure, as evaluated by the Harris-Benedict equation. Intervention group patients received a balanced diet scheme, based on a caloric intake reduction related to BMI and sex (range: 1200-1500 kcal/d for women, 1300-1600 kcal/d for men).
  Other Names: hypo-caloric diet

SUMMARY:
The relative risk of psoriasis and its severity are directly related to the body mass index (BMI).Patients with psoriasis likely undergo a vicious circle where obesity and skin disease reinforce each other. To investigate patients' opinion about their body weight (BW), the possibility of dietary approach to psoriasis, and to examine the adherence and the effects of hypo-energetic diet to maintain disease remission in obese patients a dedicated questionnaire was administered to 200 consecutive patients (125 men and 75 women) with moderate-to-severe chronic plaque psoriasis investigating whether diet factors could influence psoriasis severity and course. In second part of study, obese patients with psoriasis in remission (PASI improvement ≥ 75%) for at least 12 weeks after methotrexate therapy were randomly assigned to receive a hypo-caloric diet or free diet for 24 weeks, and then followed up for additional 12 weeks.

DETAILED DESCRIPTION:
Chronic plaque psoriasis is an inflammatory skin disease associated with obesity in 13-34% of cases. In recent years, the prevalence of overweight and obesity has increased in almost all developed countries.Obesity and a high body mass index have been shown to be risk factors for the development of psoriasis and in large, prospective studies obesity precede the development of psoriasis. More recently, obesity in adulthood has been shown to be a risk factor also for psoriatic arthritis. On the other hand, ones psoriasis has been established it may favor behaviors facilitating overweight and obesity.

To investigate patients' opinion about their BW, the possibility of dietary approach to psoriasis, a specific questionnaire was administered to 200 consecutive patients with moderate-to-severe chronic plaque psoriasis. In a second part of the study, a 24-week randomized, controlled, investigator-blinded clinical trial was performed on a limited number of patient to see whether hypo-caloric diet to maintain disease remission in obese patients previously treated with methotrexate. Patients were recruited from those consecutively admitted to the psoriasis outpatient clinic of the University Hospital of Verona. The inclusion criteria were: patients ≥ 18 year of age with moderate to severe psoriasis and a BMI ≥ 30 and without psoriasis arthritis, who were treated with methotrexate and had obtained a reduction in psoriasis severity of at least 75% (PASI 75) for the 12 weeks before enrolling into the study. Exclusion criteria were other types of psoriasis (guttate, erythrodermic and pustular psoriasis) and severe obesity (BMI >35). All patients gave their written informed consent before any study-related procedures were performed. All subjects were visited by two dermatologists who recorded demographic, biometrical, and other relevant patient's data. Visits were scheduled at screening, baseline, and every 4 weeks up to 24. Collected data included age, sex, weight, height, BMI, psoriasis duration and concomitant medications. The dermatologist who performed the PASI scoring was unaware of the randomization assignment. Patients stopped methotrexate therapy and were randomly assigned either of two groups: the first group received a low-calorie diet administered by a dietitian (intervention group) whereas the second group did not receive any dietetic recommendation (control group). Randomization was performed with the use of computer-generated random numbers and block size of 4 subjects. Patients underwent clinical and nutritional follow-up every month. The low-calorie diet was designed to achieve a loss of 5-10% of initial body weight. The caloric restriction was 500 kcal below the resting energy expenditure, as evaluated by the Harris-Benedict equation. Intervention group patients received a balanced diet scheme, based on a caloric intake reduction related to BMI and sex (range: 1200-1500 kcal/d for women, 1300-1600 kcal/d for men). Relapses were considered as loss of 50% of PASI improvement score from baseline pre-methotrexate value.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 18 year of age with moderate to severe psoriasis and a BMI ≥ 30 and without psoriasis arthritis, who were treated with methotrexate and had obtained a reduction in psoriasis severity of at least 75% (PASI 75) for the 12 weeks before enrolling into the study.
* all patients gave their written informed consent before any study-related procedures were performed.

Exclusion Criteria:

* other types of psoriasis (guttate, erythrodermic and pustular psoriasis) and severe obesity (BMI >35).
* exclusion criteria were other types of psoriasis (guttate, erythrodermic and pustular psoriasis) and severe obesity (BMI >35).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
difference in PASI at week 24 between obese psoriatic patients who underwent hypocaloric diet compared to those in free diet after obtaining a PASI reduction >75 following methotrexate. | 24 weeks

SECONDARY OUTCOMES:
patients' opinion about their body weight and it's relation with psoriasis | baseline (0 week)

CONTACTS AND LOCATIONS:
Overall Officials: Giampiero Girolomoni, Professor, Study Chair — Universita di Verona